CLINICAL TRIAL: NCT02258009
Title: A Randomized, Single-blinded, Multicenter, Phase IV Study to Compare Systemic VEGF Protein Dynamics Following Monthly Intravitreal Injections of 0.5 mg Ranibizumab Versus 2 mg Aflibercept Until Study Week 12 in Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: Systemic VEGF Protein Dynamics Following Intravitreal Injections of Ranibizumab Versus Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: TIDE DME
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002DDE25
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Visual Impairment Due to Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Monthly intravitreal injections of 0.5 mg ranibizumab
  Interventions: Drug: Ranibizumab
- Group 2 (Experimental): Three monthly intravitreal injections of 2 mg aflibercept followed by three monthly intravitreal injections of 0.5 mg ranibizumab
  Interventions: Drug: Ranibizumab; Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg intravitreal injections
  Other Names: Lucentis
Drug: Aflibercept — 2 mg intravitreal injections
  Other Names: Eylea
  Arms: Group 2

SUMMARY:
The purpose of the study is to compare the effect of intravitreal injections of ranibizumab and aflibercept on systemic VEGF protein levels in DME patients in a detailed time course.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Visual impairment predominantly due to DME.

Exclusion Criteria:

* Stroke or myocardial infarction less than 3 months prior to screening.
* Presence of uncontrolled systolic blood pressure or diastolic blood pressure
* Renal failure requiring dialysis or renal transplant or renal insufficiency
* Untreated diabetes mellitus
* Use of any systemic anti-VEGF drugs
* Use of systemic or inhaled corticosteroids for at least 30 consecutive days within 3 months prior to screening.
* Women who are pregnant or breast feeding or who are menstruating and capable of becoming pregnant* and not practicing a medically approved method of contraception

For either eye:

* Any active periocular or ocular infection or inflammation
* Uncontrolled glaucoma
* Neovascularization of the iris or neovascular glaucoma
* History of treatment with any anti-angiogenic drugs

For study eye:

* Atrophy or fibrosis involving the center of the fovea at the time of screening or baseline.
* Cataract (if causing significant visual impairment), planned cataract surgery during the study period, vitrectomy, aphakia, glaucoma surgery, severe vitreous hemorrhage, rhegmatogenous retinal detachment, proliferative retinopathy or choroidal neovascularization or macular edema of any other cause than DME
* Irreversible structural damage within 0.5 disc diameter of the center of the macula
* Panretinal laser photocoagulation within 6 months prior to randomization.
* Focal/grid laser photocoagulation within 3 months prior to randomization.
* Any intraocular procedure (including cataract surgery, Yttrium-Aluminum-Garnet capsulotomy) within 3 months prior to baseline or anticipated within the next 6 months following
* Topical ocular corticosteroids administered for at least 30 consecutive days within 3 months prior to screening.
* Application of intravitreal corticosteroids in vitreous within 6 months prior to screening. Prior application of fluocinolonacetonid releasing implant in vitreous within 36 months prior to screening.

For fellow eye

- Retinal or choroidal neovascularization or macula edema of any cause

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Systemic VEGF-A protein levels | From baseline to study week 12
  Systemic VEGF-A protein levels following monthly intravitreal injections of 0.5 mg ranibizumab versus 2 mg aflibercept (Area under the curve)

SECONDARY OUTCOMES:
Systemic VEGF-A protein levels | From study week 12 to 24
  Systemic VEGF-A protein levels in patients switching from monthly 2 mg aflibercept injections to monthly 0.5 mg ranibizumab compared to patients treated with 0.5 mg ranibizumab from baseline
Systemic VEGF-A levels | From study week 12 to 24
  Adjustment of systemic VEGF-A levels of patients switching from aflibercept to ranibizumab to levels comparable to baseline or to levels comparable as in patients treated from baseline with ranibizumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Chemnitz, Germany